CLINICAL TRIAL: NCT04335643
Title: A Remotely Delivered CBT Intervention for Youth With cSLE: A Multi-site Patient-engaged Investigation
Brief Title: Telehealth CBT for Adolescents and Young Adults With Childhood-onset Systemic Lupus Erythematosus
Acronym: cSLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Arthritis Foundation (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003882
Record Dates: First submitted 2020-02-27; First posted 2020-04-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus; depression; depressive symptoms; fatigue; pain; SLE; rheumatic disease; rheumatology; telehealth; CBT
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Depression; Fatigue; Pain; Rheumatic Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will either be randomly assigned to the intervention or to a wait-list period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEACH (Experimental): Participants will undergo CBT and continue medical TAU.
  Interventions: Behavioral: TEACH
- Control (No Intervention): Participants will only continue medical TAU.

INTERVENTIONS:
Behavioral: TEACH — TEACH is a remotely delivered psychological intervention. It consists of six one-hour weekly sessions that are HIPAA compliant and conducted over video conferencing.
  Other Names: Treatment and Education Approach for Childhood-onset Lupus
  Arms: TEACH

SUMMARY:
This study aims to investigate the feasibility and effectiveness of a remotely delivered psychological intervention for youth with cSLE. This intervention aims to teach participants skills in order to cope with fatigue, pain, and depressive symptoms--symptoms that commonly affect adolescents and young adults with lupus.

DETAILED DESCRIPTION:
This project is investigating whether a remotely delivered psychological intervention is acceptable and beneficial to teens and young adults coping with cSLE. This study uses a cognitive behavioral therapy (CBT) intervention called the Treatment and Education Approach for Childhood-onset Lupus (TEACH) to address symptoms of fatigue, depression, and pain that commonly occur in individuals with cSLE. The TEACH program includes six-weekly, one hour sessions, conducted over HIPAA-compliant video conferencing.

Participation in this study will take approximately 8-15 weeks, with a follow-up survey occurring 3-months after post-assessment, and a long-term follow-up survey occurring between 12-27 months after post-assessment. After qualifying for the study, participants will be randomly selected, like flipping a coin, to the TEACH program plus medical treatment as usual (TAU) OR medical TAU alone for six weeks. After this six-week time period, a post-assessment will be completed. Participants that only continued medical TAU will then be eligible to receive TEACH after completing the post-assessment. If these participants choose to undergo the TEACH treatment, they will be asked to complete a short interview about the program and answer questions about how their mood, pain, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with cSLE, meeting the revised American College of Rheumatology Classification Criteria for SLE by age 18 years
* Participants must have at least one elevation (based off of screening measures) in fatigue, or depressive symptoms, or pain
* Patient participants must have English language proficiency
* For participants under age 18, must have a primary caregiver willing to participate.

Exclusion Criteria:

* Patients with other chronic medical conditions (e.g., juvenile arthritis),
* Patients with a documented developmental delay, severe cognitive impairment, or thought disorder
* Patients with an untreated major psychiatric illness (e.g., bipolar disorder, psychosis, severe depression, or active suicidal ideation)
* Patients currently receiving psychological treatment for depression, fatigue or pain will be excluded to prevent overlapping treatments that may confound outcomes.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Recruitment rates of the study | After enrollment period, approximately 2 years
  Recruitment rates will be measured by the number of participants who agree to participate in the study. This information will be collected after the enrollment period.
Retention rates of the study | After data collection period, approximately 2 years
  Retention rates will be measured by the number of participants who complete the study. This information will be collected after the data collection period ends.
Feasibility of remotely-delivered TEACH | Approximately 8 weeks
  Feasibility will be measured by participant feedback in a qualitative interview.

SECONDARY OUTCOMES:
Changes in fatigue, as measured by the PROMIS Fatigue SF | Approximately 4 weeks
  The adult PROMIS Fatigue SF measures fatigue one a scale of 10-40; 10 indicating no fatigue, 40 indicating high levels of fatigue. The pediatric PROMIS Fatigue SF measures on a scale of 0-40; 0 indicating no fatigue and 40 indicating high levels of fatigue. This is to assess changes at a midpoint in the study.
Changes in fatigue, as measured by the PROMIS Fatigue SF | Approximately 8 weeks
  The adult PROMIS Fatigue SF measures fatigue one a scale of 10-40; 10 indicating no fatigue, 40 indicating high levels of fatigue. The pediatric PROMIS Fatigue SF measures on a scale of 0-40; 0 indicating no fatigue and 40 indicating high levels of fatigue.
Long-term changes in fatigue, as measured by the PROMIS Fatigue SF | Between 20 and 32 weeks, and 12-27 from post-assessment
  The adult PROMIS Fatigue SF measures fatigue one a scale of 10-40; 10 indicating no fatigue, 40 indicating high levels of fatigue. The pediatric PROMIS Fatigue SF measures on a scale of 0-40; 0 indicating no fatigue and 40 indicating high levels of fatigue.
Changes in depressive symptoms, as measured by the Children's Depression Inventory-2 (CDI-2) and Beck Depression Inventory-II (BDI-II) | Approximately 4 weeks
  The CDI-2 measures depressive symptoms on a scale of 0-54, with 0 indicating low levels of depressive symptoms, and 54 indicating high levels of depressive symptoms. The BDI-II measures depressive symptoms on a scale of 0 to 63, with 0 indicating low levels of depressive symptoms and 63 indicating high levels of depressive symptoms. This is to assess changes at a midpoint in the study.
Changes in depressive symptoms, as measured by the Children's Depression Inventory-2 (CDI-2) and Beck Depression Inventory-II (BDI-II) | Approximately 8 weeks
  The CDI-2 measures depressive symptoms on a scale of 0-54, with 0 indicating low levels of depressive symptoms, and 54 indicating high levels of depressive symptoms. The BDI-II measures depressive symptoms on a scale of 0 to 63, with 0 indicating low levels of depressive symptoms and 63 indicating high levels of depressive symptoms.
Long-term changes in depressive symptoms, as measured by the Children's Depression Inventory-2 (CDI-2) and Beck Depression Inventory-II (BDI-II) | Between 20 and 32 weeks, and 12-27 from post-assessment
  The CDI-2 measures depressive symptoms on a scale of 0-54, with 0 indicating low levels of depressive symptoms, and 54 indicating high levels of depressive symptoms. The BDI-II measures depressive symptoms on a scale of 0 to 63, with 0 indicating low levels of depressive symptoms and 63 indicating high levels of depressive symptoms.

OTHER OUTCOMES:
Changes in pain, as measured by the Pain Visual Analog Scale (VAS) | Approximately 4 weeks
  The Pain VAS measures three items on a scale of 0-10, with 0 indicating no pain and 10 indicating the worst possible pain. This is to assess changes at a midpoint in the study.
Changes in pain, as measured by the Pain Visual Analog Scale (VAS) | Approximately 8 weeks
  The Pain VAS measures three items on a scale of 0-10, with 0 indicating no pain and 10 indicating the worst possible pain
Long-term changes in pain, as measured by the Pain Visual Analog Scale (VAS) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The Pain VAS measures three items on a scale of 0-10, with 0 indicating no pain and 10 indicating the worst possible pain
The number of adverse childhood experiences, as measured by Adverse Childhood Events (ACEs) | Through study completion, up to 32 weeks, and between 12-27 months from post-assessment
  The ACEs questionnaire poses 9 different potential adverse childhood experiences in which participants indicate if they have or have not had that experience. The total is calculated by adding the items indicated as "yes."
Changes in caregivers' depression, anxiety, and stress as measured by the Depression Anxiety and Stress Scales 21 (DASS21) | Approximately 8 weeks
  The DASS21 depression, anxiety, and stress on a scale of 0-63 with 0 indicating low levels of these feelings, and 63 indicating high levels. This measure will only be completed by caregivers participating in the study.
Long-term changes in caregivers' depression, anxiety, and stress as measured by the Depression Anxiety and Stress Scales 21 (DASS21) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The DASS21 depression, anxiety, and stress on a scale of 0-63 with 0 indicating low levels of these feelings, and 63 indicating high levels. This measure will only be completed by caregivers participating in the study.
Changes in disease activity as measured by a Visual Analog Scale (VAS) | Approximately 8 weeks
  Disease activity will be measured by the physician on a VAS ranging from 0, indicating no activity, to 10 indicating high activity. This VAS used will be from the pediatric global health assessment.
Long-term changes in disease activity as measured by a Visual Analog Scale (VAS) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  Disease activity will be measured by the physician on a VAS ranging from 0, indicating no activity, to 10 indicating high activity. This VAS used will be from the pediatric global health assessment.
Changes in quality of life, as measured by the Pediatric Quality of Life (PedsQL) | Approximately 8 weeks
  The PedsQL measures quality of life in several aspects such as health, school, daily activities. Each item is reversed scored and transformed to a linear scale of 0-100, such that 100 indicates a high quality of life and 0 indicates a low quality of life
Long-term changes in quality of life, as measured by the Pediatric Quality of Life (PedsQL) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The PedsQL measures quality of life in several aspects such as health, school, daily activities. Each item is reversed scored and transformed to a linear scale of 0-100, such that 100 indicates a high quality of life and 0 indicates a low quality of life
Changes in pain interference, as measured by the PROMIS Pain Interference Short Form (SF) | Approximately 8 weeks
  The PROMIS Pain Interference SF measures how pain interferes with aspects of life, such as daily activities or family life. Scores range from 8 to 40 for adults and 0 to 32 for children, such that lower scores indicate little pain interference and high scores indicate high pain interference.
Long-term changes in pain interference, as measured by the PROMIS Pain Interference Short Form (SF) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The PROMIS Pain Interference SF measures how pain interferes with aspects of life, such as daily activities or family life. Scores range from 8 to 40 for adults and 0 to 32 for children, such that lower scores indicate little pain interference and high scores indicate high pain interference.
Changes in anxiety, as measured by the Screen for Child Anxiety Related Disorders (SCARED) and Screen for Adult Anxiety Related Disorders (SCAARED) | Approximately 8 weeks
  The SCARED measures anxiety in children on a scale of 0 to 82, such that lower scores indicates low levels of anxiety, and high scores indicated high levels of anxiety. The SCAARED measures anxiety in adults on a scale of 0 to 88 such that lower scores indicated lower levels of anxiety and high scores indicate higher levels of anxiety. Both scales are comprised of sub-scales to measure types of anxiety (such as separation anxiety).
Long-term changes in anxiety, as measured by the Screen for Child Anxiety Related Disorders (SCARED) and Screen for Adult Anxiety Related Disorders (SCAARED) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The SCARED measures anxiety in children on a scale of 0 to 82, such that lower scores indicates low levels of anxiety, and high scores indicated high levels of anxiety. The SCAARED measures anxiety in adults on a scale of 0 to 88 such that lower scores indicated lower levels of anxiety and high scores indicate higher levels of anxiety. Both scales are comprised of sub-scales to measure types of anxiety (such as separation anxiety).
Changes in disease activity, as measured by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K) | Approximately 8 weeks
  The SLEDAI 2K measures disease activity in SLE, and takes into consideration descriptors of the disease such as arthritis and vasculitis. Higher scores indicate more active disease/flares, and lower scores indicated less disease activity.
Long-term changes in disease activity, as measured by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The SLEDAI 2K measures disease activity in SLE, and takes into consideration descriptors of the disease such as arthritis and vasculitis. Higher scores indicate more active disease/flares, and lower scores indicated less disease activity.
Changes in disease activity, as measured by the Systemic Lupus International Collaborating Clinics/ACR Damage Index for Systemic Lupus Erythematosus (SLICC) | Approximately 8 weeks
  The SLICC measures disease activity by assessing descriptors in SLE. Higher scores indicate greater disease activity, lower scores indicate lesser disease activity
Long-term changes in disease activity, as measured by the Systemic Lupus International Collaborating Clinics/ACR Damage Index for Systemic Lupus Erythematosus (SLICC) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The SLICC measures disease activity by assessing descriptors in SLE. Higher scores indicate greater disease activity, lower scores indicate lesser disease activity
Changes in resilience, as measured by the Brief Resilience Scale (BRS) | Approximately 8 weeks
  The BRS measures resilience on a scale of 1 to 5 such that higher scores indicate greater resilience and lower scores indicate lower resilience.
Long-term changes in resilience, as measured by the Brief Resilience Scale (BRS) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The BRS measures resilience on a scale of 1 to 5 such that higher scores indicate greater resilience and lower scores indicate lower resilience.
Changes in medication adherence, as measured by the Medication Adherence Self-Report Inventory (MASRI) | Approximately 8 weeks
  The MASRI measures medication adherence on a scale of 0%-100%, such that lower scores indicate less adherence and higher scores indicate more adherence.
Long-term changes in medication adherence, as measured by the Medication Adherence Self-Report Inventory (MASRI) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  The MASRI measures medication adherence on a scale of 0%-100%, such that lower scores indicate less adherence and higher scores indicate more adherence.
Concomitant medications | Through study completion, up to 32 weeks, and between 12-27 months from post-assessment
  Medications will be collect through medical charts and reported by participants and caregivers of participants who are under 18 years.
Changes in COVID-related distress as measured by a Visual Analog Scale (VAS) | Approximately 8 weeks
  COVID-related distress will be measured through two items on a VAS ranging from 0-10, with 0 indicated no distress and 10 indicating extreme distress
Long-term changes in COVID-related distress as measured by a Visual Analog Scale (VAS) | Between 20 and 32 weeks, and between 12-27 months from post-assessment
  COVID-related distress will be measured through two items on a VAS ranging from 0-10, with 0 indicated no distress and 10 indicating extreme distress
Negative Treatment Effects as measured by the Negative Effects Questionnaire 20 (NEQ) | Between 8 and 32 weeks, and between 12-27 months from post-assessment
  The 20-item NEQ measures negative effects and their impact experienced from psychological treatment. The NEQ measures frequency of negative events on a scale of 0-20. If a negative event is indicated, participants are asked to indicate the severity of its impact on a scale of 0-4 with higher ratings indicating greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Natoshia Cunningham, PhD, Principal Investigator — Michigan State University
Locations (2):
- Michigan State University, Grand Rapids, Michigan, United States
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham NR, Miller A, Ely SL, Reid MR, Danguecan A, Mossad SI, Pereira LF, Abulaban K, Kessler E, Rosenwasser N, Nanda K, Rubinstein T, Reeves M, Kohut SA, Stinson J, Tal TE, Levy DM, Hiraki L, Smitherman EA, Knight AM. A multi-site pilot randomized clinical trial of the Treatment and Education Approach for Childhood-onset Lupus (TEACH) program: study design and COVID-19 adaptations. Pediatr Rheumatol Online J. 2023 Jun 23;21(1):61. doi: 10.1186/s12969-023-00835-6. PMID 37353795